CLINICAL TRIAL: NCT05500209
Title: Efficacy of Chatbot-based Internet Intervention for Stress Among University Students: A Randomized Controlled Trial
Brief Title: Chatbot-based Internet Intervention for Stress Among University Students (Stressbot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Principal Investigator, Ewelina Smoktunowicz, Principal Investigator, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stressbot
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coping Self-Efficacy (Experimental): Experimental condition enhancing coping self-efficacy
  Interventions: Behavioral: Personal resources' enhancement: self-efficacy
- Waitlist control (No Intervention): Waitlist control condition

INTERVENTIONS:
Behavioral: Personal resources' enhancement: self-efficacy — Participants in this condition are asked to take part in a 7-day psychological intervention delivered through Facebook Messenger chat-bot. Each day one CBT-framed exercise aimed at coping self-efficacy enhancement is delivered. An exercise takes form 5 to 30 minutes to complete.
  Arms: Coping Self-Efficacy

SUMMARY:
The aim of this study is to verify the efficacy of chatbot internet intervention for reduction of stress and improvement of quality of life among university students through the enhancement of coping self-efficacy.

DETAILED DESCRIPTION:
University students experience high stress levels and mental health risks. Research shows that increasing resources such as coping self-efficacy can reduce stress. Internet interventions can be successfully employed to deliver programs for improving university students' mental health.

The primary objective of this randomized controlled trial is to evaluate short- and long-term efficacy of coping self-efficacy enhancing intervention in reducing university students' stress and improving quality of life. The intervention will be delivered through a Facebook Messenger chat-bot. The secondary goal is to investigate acceptability of a chat-bot delivered intervention.

Participants will be recruited via social media and randomized to 1 of 2 groups: (1) experimental condition increasing coping self-efficacy with a 7-day program delivered through a chat-bot, or (2) waitlist control group. Outcomes include perceived stress and quality of life. Measurements will be taken at baseline (T1), immediately after intervention (T2), at 1 month follow-up (T3), and at 6 months follow-up (T4). Linear mixed effects model will be used to analyze the data.

The study aims to assess Stressbot's potential benefit for improving university students' well-being. Moreover, it will provide insight into feasibility of using chat-bots for delivering smartphone-based e-health treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* University students
* Mobile personal device with internet access

Exclusion Criteria:

* Not meeting at least 1 inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2022-11-13 (Actual)

PRIMARY OUTCOMES:
Change on Perceived Stress Scale 4 (PSS-4) | Change from baseline on PSS-4 (7 days)
  The PSS-4 is a measure of perceived stress. It consists of 4 items with response scale from 0 to 4. Higher total score represents higher perceived stress.
Change on Perceived Stress Scale 4 (PSS-4) | Change from baseline on PSS-4 (1 month)
  The PSS-4 is a measure of perceived stress. It consists of 4 items with response scale from 0 to 4. Higher total score represents higher perceived stress.
Change on Perceived Stress Scale 4 (PSS-4) | Change from baseline on PSS-4 (6 month)
  The PSS-4 is a measure of perceived stress. It consists of 4 items with response scale from 1 to 4. Higher total score represents higher perceived stress.
Change on Brunnsviken Brief Quality of Life Scale (BBQ) | Change from baseline on BBQ (7 days)
  The BBQ is a measure of quality of life. It consists of 12 items with response scale from 0 to 4. Higher total score represents higher quality of life.
Change on Brunnsviken Brief Quality of Life Scale (BBQ) | Change from baseline on BBQ (1 month)
  The BBQ is a measure of quality of life. It consists of 12 items with response scale from 0 to 4. Higher total score represents higher quality of life.
Change on Brunnsviken Brief Quality of Life Scale (BBQ) | Change from baseline on BBQ (6 months)
  The BBQ is a measure of quality of life. It consists of 12 items with response scale from 0 to 4. Higher total score represents higher quality of life.

SECONDARY OUTCOMES:
Coping Self-Efficacy Scale (CSES) | Change from baseline on CSES (7 days)
  The CSES is a measure of coping self-efficacy. It consists of 26 items with response scale from 1 to 10. Higher total score represents higher coping self-efficacy.
Coping Self-Efficacy Scale (CSES) | Change from baseline on CSES (1 month)
  The CSES is a measure of coping self-efficacy. It consists of 26 items with response scale from 1 to 10. Higher total score represents higher coping self-efficacy.
Coping Self-Efficacy Scale (CSES) | Change from baseline on CSES (6 months)
  The CSES is a measure of coping self-efficacy. It consists of 26 items with response scale from 1 to 10. Higher total score represents higher coping self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Ewelina Smoktunowicz, PhD, Principal Investigator — 1Department of Psychology, SWPS University of Social Sciences and Humanities, Warsaw, Poland
Locations (1):
- SWPS University of Social Sciences and Humanities, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakker D, Kazantzis N, Rickwood D, Rickard N. A randomized controlled trial of three smartphone apps for enhancing public mental health. Behav Res Ther. 2018 Oct;109:75-83. doi: 10.1016/j.brat.2018.08.003. Epub 2018 Aug 11. PMID 30125790
- [Background] Hobfoll SE. Conservation of resources. A new attempt at conceptualizing stress. Am Psychol. 1989 Mar;44(3):513-24. doi: 10.1037//0003-066x.44.3.513. PMID 2648906
- [Background] Amanvermez Y, Zhao R, Cuijpers P, de Wit LM, Ebert DD, Kessler RC, Bruffaerts R, Karyotaki E. Effects of self-guided stress management interventions in college students: A systematic review and meta-analysis. Internet Interv. 2022 Feb 12;28:100503. doi: 10.1016/j.invent.2022.100503. eCollection 2022 Apr. PMID 35242591
- [Background] Smoktunowicz E, Lesnierowska M, Carlbring P, Andersson G, Cieslak R. Resource-Based Internet Intervention (Med-Stress) to Improve Well-Being Among Medical Professionals: Randomized Controlled Trial. J Med Internet Res. 2021 Jan 11;23(1):e21445. doi: 10.2196/21445. PMID 33427674